CLINICAL TRIAL: NCT00002437
Title: A Phase II/III Study of the Safety and Efficacy of 1-(S)-(3-Hydroxy-2-Phosphonylmethoxypropyl)Cytosine Dihydrate (Cidofovir; HPMPC) for the Treatment of Peripheral Cytomegalovirus Retinitis in Patients With AIDS
Brief Title: The Safety and Effectiveness of Cidofovir in the Treatment of Cytomegalovirus (CMV) of the Eyes in Patients With AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 216A; GS-93-106
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-11

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Probenecid; Drug Therapy, Combination; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents; cidofovir
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Cidofovir; Probenecid

INTERVENTIONS:
Drug: Cidofovir
Drug: Probenecid

SUMMARY:
To determine whether cidofovir (HPMPC) therapy administered by intravenous infusion can extend the time to progression of peripheral cytomegalovirus (CMV) retinitis in AIDS patients. To evaluate the safety and tolerance of HPMPC therapy when administered by intravenous infusion in AIDS patients with CMV retinitis that is not immediately sight-threatening. To evaluate the virologic effects of intravenous HPMPC therapy on CMV shedding in urine, blood, and/or semen. To evaluate the impact of HPMPC therapy on visual acuity.

DETAILED DESCRIPTION:
Patients are randomized to one of two treatment arms. Group A receives HPMPC by IV infusion weekly for 2 consecutive weeks (induction) and then every other week (maintenance) with oral probenecid and IV hydration. Group B receives no treatment until the time of retinitis progression (deferred treatment), at which time they receive the same regimen as Group A, provided retinitis progression is not immediately sight-threatening.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral agents.
* Oral trimethoprim/sulfamethoxazole.
* Aerosolized pentamidine.
* Dapsone.
* Fluconazole.
* Rifabutin.
* Filgrastim (G-CSF).
* p24 vaccine.

Patients must have:

* Diagnosis of AIDS by CDC criteria.
* Diagnosis of peripheral (not immediately sight-threatening) CMV retinitis.
* Visual acuity in the affected eye of >= three lines on the ETDRS (Early Treatment Diabetic Retinopathy Study) chart at 1 m distance.
* Life expectancy of at least 3 months.
* Consent of parent or guardian in patients less than 18 years of age.

Prior Medication:

Allowed:

* Acyclovir.
* Prior ganciclovir, foscarnet, or CMV hyperimmune immunoglobulin if given solely as prophylaxis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Media opacity that precludes visualization of the fundus of both eyes.
* Retinal detachment.
* Clinically significant cardiac disease, including symptoms of ischemia, congestive heart failure, or arrhythmia.
* Active medical problems considered sufficient to hinder study compliance.
* Known clinically significant allergy to probenecid.

Concurrent Medication:

Excluded:

* Acyclovir (may be reinstituted following development of herpetic lesions).
* Ganciclovir.
* Foscarnet.
* Amphotericin B.
* Diuretics.
* Aminoglycoside antibiotics.
* CMV hyperimmune immunoglobulin.
* Intravenous pentamidine.
* Other nephrotoxic agents.
* Other investigational drugs with potential nephrotoxicity.

Prior Medication:

Excluded:

* Prior ganciclovir, foscarnet, or CMV hyperimmune immunoglobulin as therapy for CMV disease (although permitted if previously received solely as prophylaxis).

Excluded within 1 week prior to study entry:

* Amphotericin B.
* Vidarabine.
* Other nephrotoxic agents.
* Aminoglycoside antibiotics.
* Intravenous pentamidine. Drug or alcohol abuse.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - Mount Zion Med Ctr, San Francisco, California
  - Beth Israel Hosp, Boston, Massachusetts
  - Besselaar Associates, Princeton, New Jersey
  - Univ of Rochester Med Ctr, Rochester, New York
  - Univ of North Carolina Hosps, Chapel Hill, North Carolina
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
- Charing Cross and Westminster Med School, London Southwest 10, United Kingdom

REFERENCES:
- [Background] Lalezari J, et al. A phase II/III randomized study of immediate versus deferred intravenous (IV) cidofovir (CDV, HPMPC) for the treatment of peripheral CMV retinitis (CMV-R) in patients with AIDS. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:170